CLINICAL TRIAL: NCT04951947
Title: A Prospective, Single-arm Phase II Clinical Study to Evaluate the Efficacy and Safety of JS-201 Combined With Lenvatinib in the Treatment of Small-cell Lung Cancer With Previous Chemotherapy Combined With PD-L1 Failure
Brief Title: JS-201 Combined With Lenvatinib in the Treatment of Small-cell Lung Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Yongchang Zhang, Director, Head of Medical Oncology, Principal Investigator, Clinical Professor, Hunan Province Tumor Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS-201
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Small-cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm A (Experimental): Treatment arm
  Interventions: Drug: JS201 combine with Lenvatinib

INTERVENTIONS:
Drug: JS201 combine with Lenvatinib — JS201 300mg i.v Q2wLenvatinib 8mg po. Qd

SUMMARY:
This is a prospective, single-arm phase II clinical study to evaluate the efficacy and safety of JS-201 combined with lenvatinib in the treatment of small-cell lung cancer that has failed previous chemotherapy combined with PD-L1. The primary observational endpoint is ORR, and the secondary observational endpoint is PFS, OS. The intervention mode is JS201 300mg i.v Q2w, lenvatinib 8mg po. Qd.

ELIGIBILITY:
Inclusion Criteria:

* 1. The imaging diagnosis is the extensive stage of SCLC
* 2. The patient failed first-line EC+PD-L1 treatment
* 3 PS 0-1

Exclusion Criteria:

* 1. Diagnosed as non-small cell lung cancer
* 2. Women during pregnancy
* 3. Patients with symptomatic brain metastases
* 4. PS≥2

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 1 year
  Defined as the proportion of subjects in complete remission (CR) and partial remission (PR) to the total subjects

SECONDARY OUTCOMES:
PFS | 1 year
  Defined as the time from the beginning of treatment to the first imaging disease progression or death (whichever occurs first)

CONTACTS AND LOCATIONS:
Overall Officials: Yongchang Zhang, MD, Principal Investigator — Hunan Cancer Hospital
Locations (1):
- Hunan Cancer Hospital, Changsha, Hunan, China